CLINICAL TRIAL: NCT01616667
Title: Posterior Approach Versus Lateral Approach in Osteoarthritis Patients, With Primary Total Hip Arthroplasty. The Effect on Early Physical Function, Pain, Patient Reported Outcome Measures, Gait and Muscle Weakness A Randomized Clinical Trial
Brief Title: Comparing the Clinical Effects of Posterior Approach Versus Lateral Approach in Osteoarthritis Patients With a THA
Acronym: COMPALA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Orthopaedic department of Køge Hospital (Unknown); Region Zealand (Other); Region of Southern Denmark (Other); University of Southern Denmark (Other); The Danish Rheumatism Association (Other); Bevica Fonden (Other); Bjarne Jensens Fond (Unknown)
Responsible Party: Principal Investigator, Signe Rosenlund, MD, ph.d. student, MD, ph.d.-student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-20120009; A2116 Signe Rosenlund (Other: The Danish Rheumatism Association); 11/28589 (Other: Region of Southern Denmark)
Record Dates: First submitted 2012-05-30; First posted 2012-06-12 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Unilateral Primary Osteoarthritis of Hip
Keywords: Controlled Clinical Trial; Operative Surgical Procedures; Treatment Outcome; Pain Measurement; Quality of Life; Questionnaires/standards; Activities of Daily Living; Biomechanics; Gait*; Hip Joint/physiology*; Hip Joint/surgery*; Recovery of Function/physiology
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified direct lateral approach (Active Comparator): The patients included is operated with a total hip arthroplasty using a modified direct lateral approach
  Interventions: Procedure: Total hip arthroplasty
- Posterior approach (Active Comparator): The patients included is operated with a total hip arthroplasty using posterior approach
  Interventions: Procedure: Total hip arthroplasty

INTERVENTIONS:
Procedure: Total hip arthroplasty — The patients included is operated with a total hip arthroplasty due to primary osteoarthritis

SUMMARY:
The aim of this study is to investigate the clinical outcome of the two different, but widely used, surgical approaches (Posterior approach and Lateral approach) of primary total hip arthroplasty in patients diagnosed with osteoarthritis. This study is divided into one main study and two sub-studies. The main study investigates the patient-reported outcome measures (questionnaire) within the first year post surgery. The two sub-studies investigate; i) the level of physical function and pain within the first 3 month after surgery, and ii) investigate the potential difference the two approaches have on gait-patterns and maximal isometric hip-muscle-strength, within the first year after surgery. Both approaches are described with potential drawbacks. Posterior approach has a higher risk of dislocation of the prostheses and revision due to dislocation compared with Lateral approach. Contrary, Lateral approach is described with the potential drawbacks of pain, lower physical function, gait abnormalities and muscle weakness, leading to less satisfied patients. However, according to a Cochrane analysis from 2004 concludes, more investigation is needed to determine the extent of differences.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45-70 years, both included.
* Patients schedule for primary cementless total hip arthroplasty.
* Endstage hip osteoarthritis(OA) or minor dysplasia of the hip(CE-angle > 20 degrees).

Exclusion Criteria:

1. more major joint (hip or knee) than the current hip affected with OA, with expected joint replacement surgery within a year.
2. Prior joint replacement surgery on any major joint (hip, knee) in lower limb.
3. BMI above 35.
4. Any physical disability that prevents patients from walking 20 meters without aid.
5. The patients is not suitable for standard cementless prosthetic components.
6. Any neurological disease (ex. cerebral thrombosis, Parkinson) compromising the walking ability.
7. Any severe medical condition compromising walking ability (ex. chronic heart failure, chronic obstructive pulmonary disease).
8. Severe dementia.
9. Inability to read and understand Danish writing and oral instructions.
10. Do not want to participate

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Hip Disability and Osteoarthritis Outcome Score (HOOS)-Physical Function Short form(HOOS-PS), 12 month | Endpoint 12 month
  Primary study:
  Hip Disability and Osteoarthritis Outcome Score (HOOS) includes five subscales: 1)Pain 2) Other symptoms 3) Activities of daily living(ADL) 4) Sport and recreation function and 5) Hip related quality of life. HOOS-Physical Function Short form (HOOS-PS) is an aggregation and shortening of the two original subscales of HOOS-ADL and Sport and Recreation. HOOS-PS is a validated instrument. HOOS has been translated to Danish.
  We will use HOOS-PS as primary outcome.

SECONDARY OUTCOMES:
Hip Disability and Osteoarthritis Outcome Score (HOOS)-pain, 12 month | Baseline, 3 month, 6 month and endpoint 12 month
  Primary study
Hip Disability and Osteoarthritis Outcome Score (HOOS)-Hip related quality of life, 12 month | Baseline, 3 month, 6 month and endpoint 12 month
  Primary study
University of California Los Angeles activity score (UCLA), 12 month | Baseline, 3 month, 6 month and endpoint 12 month
  Primary study:
  University of California Los Angeles activity score (UCLA) is a score focusing on patient activity level. The score is based on a scale from 1 to 10, ranging from inactive to regularly participate in impact sport or heavy labor. UCLA contributes with important qualitative information with regard to patient activity in correlation with other clinical outcome measures. UCLA is found reliable and valid and is translated to Danish.
EQ-5D self-rated health index -and EQ VAS scores, 12 month | Baseline, 3 month, 6 month and endpoint 12 month
  Primary study:
  EuroQol/EQ-5D is a standardized, reliable and validated instrument to measure quality of life. The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and the EQ VAS that records the respondent's overall self-rated health on a vertical, visual analogue scale. EQ-5D is translated to Danish.
The 20 meter walk-test (20MeWa) | Baseline, 3 days, 21 days and endpoint 3 month
  Sub-study 1:
  The 20 meter walk-test (20MeWa). Patients are instructed to walk 20 meters between two clearly visible lines marked on the floor. The patients are instructed to walk with their usual pace on two trials and on the two following trials to walk at maximal pace, at which they feel secure. The mean velocity of each two trials are used for further analysis.
"Timed Up and Go"- test (TUG), 3 month | Baseline, 3 days, 21 days and endpoint 3 month
  Sub-study 1:
  The "Timed Up and Go" test (TUG) measures the time it takes a person to rise from a chair walk 3 meters, turn and walk back to the chair and sit down again. TUG is found to be a reliable and valid test for quantifying functional mobility.
"Repeated chair rise"- test (RCR), 3 month | Baseline, 3 days, 21 days and endpoint 3 month
  Sub-study 1:
  "Repeated chair rise"- test (RCR) assess the strength of the lower limb muscles overall. The test measures the maximum "stand and sit" cycles the test-person can perform on a chair within in 30 seconds. The test has been showed to gives a reliable and valid measurement of lower body strength in generally active older adults.
30 seconds maximal repeated unilateral knee bending, 3 month | Baseline, 3 days, 21 days and endpoint 3 month
  Sub-study 1:
  30 seconds maximal repeated unilateral knee bending. It evaluates the maximum number of knee bends performed on one leg in 30 seconds and the ability to execute fast coupled eccentric-concentric muscle force over the knee joint. The patient stand aligned with the front of their foot touching a straight line taped to the floor; finger tip support for balance is provided by the examiner. The patient is then asked to bend the knee, without bending forward from the hip, until he/she could no longer see the line at the toes (about 30º of knee flexion).
Opioid consumption, 3 month | Baseline, 1,2,3,4,5 days, 2, 3, 4, 6,8,10 weeks and endpoint 12 week
  Sub-study 1:
  The opioid consumption will be patient administrated and recorded each day, the first 5 days after surgery. After discharged the patient will fill in a patients-diary, where the analgesics consumption are registered.
Self-reported pain on a numerical ranking scale(NRS), 3 month | Baseline, 1,2,3,4,5 days, 2, 3, 4, 6,8,10 weeks and endpoint 12 week
  Sub-study 1:
  The self-reported pain on a numerical ranking scale(NRS)will be recorded each day, the first 5 days after surgery. After discharged the patient will fill in a patients-diary, where the NRS are registered.
Hip Disability and Osteoarthritis Outcome Score (HOOS)-pain, 3 month | Baseline, 5 days, 2, 3, 4, 6,8,10 weeks and endpoint 12 week
  Sub-study 1:
  We will use the Hip Disability and Osteoarthritis Outcome Score (HOOS)subscales -Pain.
  It will be recorded after discharged in a patients-diary
Hip Range of motion (ROM), 3 month | Baseline and endpoint 3 month
  Sub-study 1:
  Range of motion in the hip joint evaluated by goniometer at baseline and 3 month post-surgery Extension/Flexion. Abduction/adduction. Internal/external rotation.
Gait Deviation Index(GDI), 12 month | Baseline, 3 month, and endpoint 12 month
  Sub-study 2:
  Data from 3 dimensional gait analysis(6 camara Vicon MX Motion Analysis system), including EMG analysis during gait.
  Gait Deviation Index (GDI) was created to present gaitanalysis data in one score to give a comprehensive evaluation of the patients ambulation compared to healthy subjects. GDI is calculated from 15 kinematic variables, representing 98% of the variation in gait-patterns. A GDI score upon 100 represent normal gait. Every 10 points below this represent 1 standard deviation (SD) from normal gait.
Kinematic gait data, 12 month | Baseline, 3 month, and endpoint 12 month
  Sub-study 2:
  Data from 3 dimensional gait analysis(6 camara Vicon MX Motion Analysis system), including EMG analysis during gait.
  Kinematic:
  Sagittal hip Range of motion: extension/flexion. Frontal hip Range of motion: abduction/adduction. Frontal trunk inclination: left and right movement of the trunk.
Temporospatial parameters, 12 month | Baseline, 3 month, and endpoint 12 month
  Sub-study 2:
  Data from 3 dimensional gait analysis(6 camara Vicon MX Motion Analysis system), including EMG analysis during gait.
  Temporospatial parameters:
  Velocity. Cadance. Step duration. Stance duration
Electromyography (EMG) during walk, 12 month | Baseline, 3 month, and endpoint 12 month
  Sub-study 2:
  Data from 3 dimensional gait analysis(6 camara Vicon MX Motion Analysis system), including EMG analysis during gait.
  Electromyography (EMG)during walk:
  Peak EMG- in stance phase (absolute/normalized to MVC) Mean EMG- in stance phase (absolute/normalized to MVC) Integrated EMG during stancephase
Isometric maximal voluntary muscle contraction(MVC), 12 month | Baseline, 3 month, and endpoint 12 month
  Sub-study 2:
  Data from: Isometric maximal voluntary muscle contraction(MVC), including EMG analysis during test.
  Maximal force (Fmax):
  Hip Extension Flexion and Abduction. Rate of force development(RFD): Hip Extension. Flexion and Abduction
Limping question from Harris Hip Score | Baseline, 3 month, 6 month and endpoint 12 month
  Primary study

CONTACTS AND LOCATIONS:
Overall Officials: Signe Rosenlund, MD, Principal Investigator — Odense University Hospital and University of Southern Denmark; Søren Overgaard, MD, Professor, Study Chair — Odense University Hospital and University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Rosenlund S, Broeng L, Overgaard S, Jensen C, Holsgaard-Larsen A. The efficacy of modified direct lateral versus posterior approach on gait function and hip muscle strength after primary total hip arthroplasty at 12months follow-up. An explorative randomised controlled trial. Clin Biomech (Bristol). 2016 Nov;39:91-99. doi: 10.1016/j.clinbiomech.2016.09.011. Epub 2016 Sep 30. PMID 27721093
- [Derived] Rosenlund S, Broeng L, Jensen C, Holsgaard-Larsen A, Overgaard S. The effect of posterior and lateral approach on patient-reported outcome measures and physical function in patients with osteoarthritis, undergoing total hip replacement: a randomised controlled trial protocol. BMC Musculoskelet Disord. 2014 Oct 27;15:354. doi: 10.1186/1471-2474-15-354. PMID 25345483